CLINICAL TRIAL: NCT00306722
Title: A Phase 3, Randomized, Double-Blind, Dose-Controlled Study To Assess The Efficacy And Safety Of AQUAVAN® (Fospropofol Disodium) Injection For Minimal-To-Moderate Sedation In Patients Undergoing Flexible Bronchoscopy
Brief Title: An Effectiveness and Safety Study of AQUAVAN® Injection (Fospropofol Disodium) for Sedation During Flexible Bronchoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3000-0524; MGI 3000-0524
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Bronchoscopy; Anesthesia
Keywords: Bronchoscopy; Sedation; AQUAVAN; fospropofol disodium; Flexible bronchoscopy
MeSH Terms: interventions — fospropofol; Injections

INTERVENTIONS:
Drug: AQUAVAN® (fospropofol disodium) Injection

SUMMARY:
Very often patients receive medication before a diagnostic, therapeutic, or surgical procedure to help them relax, keep them calm, and to relieve them from pain. This is called procedural sedation. During procedural (mild-to-moderate) sedation, a patient is first given a pain-relief medication (analgesic) and then a medication to help him/her relax and keep him/her calm (sedative). Propofol is the drug commonly used for sedation because it releases immediately into the blood stream and causes fast sedation. AQUAVAN (fospropofol disodium) is made as a slow release version of propofol with a longer duration of effect.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, dose-controlled study designed to evaluate the efficacy and safety of AQUAVAN 6.5 mg/kg compared to a minimally effective dose of AQUAVAN 2.0 mg/kg, both following pretreatment with an analgesic, fentanyl in patients who are undergoing flexible bronchoscopy.

Following completion of preprocedure assessments, patients will be randomly assigned to 1 of 2 treatment groups at a 2:3 (AQUAVAN initial dose 1 [2.0 mg/kg]:AQUAVAN initial dose 2 [6.5 mg/kg] allocation ratio on the day of the scheduled procedure. Randomization will be stratified by site.

A person skilled in airway management (such as a respiratory therapist, a study nurse, or a clinician) and authorized by the facility in which the colonoscopy is performed must be immediately available during the conduct of the study. All patients will be placed on supplemental oxygen via nasal cannula (4 L/min), and an ECG monitor, pulse oximeter, and blood pressure monitor will be attached prior to administration of study medication. All patients will receive analgesic pretreatment (fentanyl citrate injection for pain; lidocaine for topical anesthetic followed by the administration of study medication. Assessments will be made to evaluate the patients for levels of sedation, clinical benefit of sedation, and adverse events. Blood samples will be collected for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand, either orally or in writing, and be able to consent and complete the required assessments and procedures
2. Patient provides signed/dated Informed Consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization after receiving a full explanation of the extent and nature of the study.
3. Patient must be at least 18 years of age at the time of screening.
4. If female, patient must be surgically sterile, postmenopausal, or not pregnant or lactating and must have been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and predose.
5. Patient meets American Society of Anesthesiologists (ASA) Physical Classification System status of P1 to P4.

Exclusion Criteria:

1. Patient has a history of allergic reaction or hypersensitivity to any anesthetic agent or opioid.
2. Patient does not meet nils per os (NPO) status per ASA guidelines or institution's guideline.
3. Patient has a Mallampati Classification Score of 4; OR a Mallampati Classification Score of 3 AND a thyromental distance ≤4 cm, or for any other reason has a difficult airway, in the opinion of the Investigator.
4. Patient has an abnormal, clinically significant 3-lead ECG finding at predosing period Day 0.
5. Patient has participated in an investigational drug study within 1 month prior to study start.
6. Patient is unwilling to adhere to pre- and postprocedural instructions.
7. Patient for whom the use of fentanyl citrate injection (fentanyl) is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Sedation Success rate is defined as: Having 3 consecutive Modified Observer's Assessment of Alertness/Sedation (OAA/S) scale scores of ≤4 after administration of sedative medication
Completing the procedure
Without requiring the use of alternative sedative medication
Without requiring manual or mechanical ventilation

SECONDARY OUTCOMES:
Treatment Success rate - Treatment Success is defined as a patient (i) completing the procedure (ii) without requiring alternative sedative medications AND (iii) without requiring manual or mechanical ventilation
Proportion of patients willing to be treated again with the same study sedative medication
Proportion of patients who do not recall being awake during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD, PharmD, Study Director — Eisai Inc.
Locations (25):
- United States (25):
  - Pulmonary Associates of Mobile, PC, Mobile, Alabama
  - Precision Trials, Phoenix, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - USC Health Science Campus (USC University Hospital), Los Angeles, California
  - Pensacola Research Consultants, Inc., Pensacola, Florida
  - Acute Care Consultants Inc., Augusta, Georgia
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Central Maine Pulmonary Associates, Auburn, Maine
  - Berkshire Medical Center, Pittsfield, Maryland
  - Hurley Medical Center, Flint, Michigan
  - Keith Popovich, MD, PLLC, Butte, Montana
  - International Heart Institue of MT Foundation, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - United Health Scrvices Hosptial, INC, Johnson City, New York
  - Brody School of Medicine, Greenville, North Carolina
  - ALL-TRIALS Clinical Research, LLC, Winston-Salem, North Carolina
  - University of Cincinnati, The University Hospital, Cincinnati, Ohio
  - Lowcountry Lung & Critical Care, PA, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - The University of Texas Medical Branch Division of APICS, Galveston, Texas
  - Johnston Memorial Hospital Pulmonary Research, Abingdon, Virginia
  - Pulmonary Associates of Fredericksburg, Inc., Fredericksburg, Virginia

REFERENCES:
- [Derived] Silvestri GA, Vincent BD, Wahidi MM, Robinette E, Hansbrough JR, Downie GH. A phase 3, randomized, double-blind study to assess the efficacy and safety of fospropofol disodium injection for moderate sedation in patients undergoing flexible bronchoscopy. Chest. 2009 Jan;135(1):41-47. doi: 10.1378/chest.08-0623. Epub 2008 Jul 18. PMID 18641105